CLINICAL TRIAL: NCT03791671
Title: Individual Balance Training vs. Group Balance Training to Improve Walking Speed Post Stroke - a Randomized, Controled Pilot Study
Brief Title: Balance Training After Stroke - a Randomized, Controled Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RehaClinic AG (Other)
Responsible Party: Principal Investigator, Mrs. Wiebke Weigert, Principal investigator, RehaClinic AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01700
Record Dates: First submitted 2018-12-20; First posted 2019-01-03 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: Balance training; Gait Speed
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: There will be a intervention group and a control group. Both groups do active treatment. In the intervention group they will have individual balance training and in the control group they will have balance training in a group from 3-6 persons. But both groups will do the same balance program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- individual balance training (Experimental): After the initial assessments, the three week intervention time begins, which is completed with the reassessments.
  The patients receive 2x weekly individual balance training for 25 minutes each. This runs in addition to the normal, prescribed rehabilitation program. The rehabilitation program includes at least 3 therapies daily. These may be group therapies, speech therapy, occupational therapy, neuropsychology and physiotherapy adapted to the needs of the patient. In physiotherapy and occupational therapy no balance training will be performed during the intervention period.
  Interventions: Other: individual balance training
- group balance training (Active Comparator): The patients receive 2x weekly group balance training for 25 minutes each. This runs in addition to the normal, prescribed rehab program. The rehabilitation program includes at least 3 therapies daily. These may be group therapies, speech therapy, occupational therapy, neuropsychology and physiotherapy adapted to the needs of the patient. In physiotherapy and occupational therapy no balance training will be performed during the intervention period.
  In group therapy are 3 to 6 patients with different neurological diagnoses. As it is usual in rehabilitation everyday life.
  Interventions: Other: group balance training

INTERVENTIONS:
Other: individual balance training — One physiotherapist trains one Patient nearby a bar. The tasks changes in gage, visual feedback, vestibular feedback and underground. The Positions will be hodl for 10-30 seconds.
  Arms: individual balance training
Other: group balance training — Like the individual balance training
  Arms: group balance training

SUMMARY:
This pilot study is part of a master's thesis. In the rehabilitation of stroke patients should be compared whether individual balance training has a greater effect than group balance training. The result is determined based on the walking speed.

DETAILED DESCRIPTION:
The RehaClinic Kilchberg is a neurological rehabilitation facility with the phases B-D. Between February and the end of March, out of 78 patients, 71% of the patients had a stroke. Therefore, my choice of topic for the Master's thesis fell on balance training of patients after a stroke. The duration of the study is based on the timetable for the Master's thesis. Initially, 20 stroke patients will be recruited. When the number is reached, the study is completed to begin descriptive statistics and analyze potential BIAS.

Deficits in the vestibular, visual, motor, and / or somatosensory systems lead to falls in the first 6 months after the stroke. This affects approximately 46% of patients. But also cognitive processes, such as attention and concentration. Therefore, the treatment must be adapted to the respective strategy of the patient. If the patient increasingly uses the visual system, the therapy has to work a lot with the eyes closed. In turn, if he uses more of the sensorimotor system is increasingly trained with unstable documents. After this system, the balance program was set up. It is the same for the intervention and control group to make a difference between individual and group training.

ELIGIBILITY:
Inclusion Criteria:

* stroke starting from Rehabilitation phase B
* ability to understand therapy instructions
* walkable with aids

Exclusion Criteria:

* Neurodegenerative disease
* non-stroke dizziness
* cardiopulmonary insufficiency
* polyneuropathy
* peripheral vascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change of the walking speed at three weeks | Measurement one day before and one day after the three weeks intervention time, Data analysis through study completion
  10m walking test

SECONDARY OUTCOMES:
Change of the balance score at three weeks | Measurement one day before and one day after the three weeks intervention time, Data analysis through study completion
  The Berg Balance Scale is used to determine the risk of falling. The BBS detects deficits at both activity and body function levels. It consists of 14 items. Some items require that the patient maintains positions of increasing difficulty, from sitting to standing on one leg. Other items evaluate the ability to perform specific tasks, such as reaching forward, turning around and picking up an object from the floor. Scoring is based on the ability to meet certain time or distance requirements and to perform the items independently. Scaling takes place from 0 points (not possible) to 4 points (independently possible). This results in a total score of 56 points. The cut-off is at 45 points.
Change of the Walking ability (walking aid) at three weeks | Measurement one day before and one day after the three weeks intervention time, Data analysis through study completion
  Functional Ambulation categories - is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device. To use the FAC, an assessor asks the subject various questions and briefly observes their walking ability to provide a rating from 0 to 5. A score of 0 indicates that the patient is a non-functional ambulator (cannot walk); A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3). A score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score).

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Teuschl, Ass.-Prof., Study Chair — Donauuniversität Krems (Danube University)
Locations (1):
- RehaClinic Kilchberg, Kilchberg, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: RehaClinic AG — http://www.rehaclinic.ch

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03791671/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT03791671/ICF_001.pdf